CLINICAL TRIAL: NCT00677560
Title: Impulse Oscillometry and Airway Inflammation in Asthma and Chronic Obstructive Pulmonary Disease and Airways Physiology in Other Lung Conditions and Healthy Lungs
Brief Title: The Natural History of Small Airways Physiology in Diseased and Healthy States
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 08/H0709/2
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-11

CONDITIONS: Asthma; COPD; Interstitial Lung Disease; Cystic Fibrosis; Patients Requiring Lung Transplant
Keywords: resistance; reactance; inflammation; lung function; respiratory function
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Cystic Fibrosis; Inflammation; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- 3: Mild-moderate asthma.
  Within the asthma group, there were two sub-groups; mild-moderate asthma and severe asthma distinguished using the Global Initiative for Asthma (GINA) guidelines (GINA, 2009).
- 4: Severe Asthma
  Within the asthma group, there were two sub-groups; mild-moderate asthma and severe asthma distinguished using the Global Initiative for Asthma (GINA) guidelines (GINA, 2009).
- 1: Normal subjects
  Normal subjects were a group made up of healthy subjects, with normal lung function, non-smokers at the time of the screening.
- 2: Healthy smokers
  Healthy smokers were comprised of people who were current smokers and had normal lung function at the time of screening.
- 5: COPD (Gold stage I - III)
  The COPD group included stage I to III patients, classified according to severity of airflow limitation (post bronchodilator FEV1), from the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (GOLD, 2011).

SUMMARY:
Spirometry is a useful clinical tool for the assessment and monitoring of lung disease, however, it does not provide information on peripheral airways resistance. On the contrary, impulse oscillometry (IOS) may provide information not only on airway resistance (Rrs) but also on the elastic properties of the lung (Xrs). In addition, multiple breath nitrogen washout (MBNW) utilizes the exhalation of nitrogen gas from the airways to determine changes in lung ventilation and derive small airways indices (that tells us about small airways calibre). This method, like IOS, allows a precise assessment of small airways function.

Even though patients with asthma may show some reduction of the caliber of the small airways these changes are more a feature of patients with COPD. The study team hypothesize that IOS and MBNW measurements may detect these differences and provide different resistance profiles for asthma and COPD. Furthermore, the study team would like to investigate the relationship between airway inflammation and small airway disease by measuring exhaled nitric oxide (NO) at multiple exhalation flow rates. This technique allows the partitioning of NO produced in the central airways from that generated more peripherally in the lung, providing valuable information on the activity of inflammation in different parts of the respiratory system. The study team hope that the combined use of IOS, MBNW and NO will identify a possible correlation between inflammation and small airway dysfunction.

DETAILED DESCRIPTION:
Background

The main objective of this study is to measure the damage of the small airways in lung disease exploring the "silent zone" with methods that have not been used before together in the same patients. Furthermore, because this is a 4 year longitudinal study, the study team will investigate the time related changes of small airway function in lung disease and normal healthy subjects.

The study will also investigate the relationship between small airway resistance and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged between 18-85 years;
* volunteers who are able to give written informed consent Patients meeting the diagnostic criteria for asthma, COPD, ILD, CF, chronic cough.

Exclusion Criteria:

* upper respiratory tract infection within the previous 28 days
* any history or evidence of renal, cardiovascular, gastrointestinal or hepatic disease
* any history and evidence of neuropsychiatric disease
* treatment with antibiotics within 4 weeks prior to the study
* alcohol, drug abuse or any other condition associated with poor compliance
* breast feeding
* pregnancy
* are unable to provide written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients will be recruited from outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2010-06-22 (Actual); Primary Completion 2013-07-10 (Actual); Study Completion 2013-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Paredi, MD, PhD, Study Director — Airway Disease Section, National Heart and Lung Institute, Imperial College, London; Omar A Usmani, MD, PhD, Principal Investigator — Airway Disease Section, National Heart and Lung Institute, Imperial College, London; Peter J Barnes, Prof, Study Chair — Airway Disease Section, National Heart and Lung Institute, Imperial College, London; Neil Pride, Prof, Study Chair — Airway Disease Section, National Heart and Lung Institute, Imperial College, London; Michael Goldman, Prof, Study Chair — Airway Disease Section, National Heart and Lung Institute, Imperial College, London
Locations (1):
- Airway Disease Section, National Heart and Lung Institute, Imperial College, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single centre cross-sectional and longitudinal study involving asthmatic and chronic obstructive pulmonary disease (COPD) patients and healthy volunteers (including smokers).
  Subjects were between the ages of 18-85 years old, were given a patient information sheet and provided their written informed consent. Subjects were interviewed at visit 1 and a medical history was documented.
Groups:
- Mild-moderate Asthma; Severe Asthma: Asthmatics (mild, moderate and severe) were classified according to the Global Initiative for Asthma diagnostic criteria (GINA, 2009).
- Normal Subjects: This group consisted of 29 never-smokers with no history of respiratory disease.
- Healthy Smokers: Healthy smokers had no history of respiratory disease, and were all current smokers
- COPD (Gold Stage I - III): COPD patients (stages I - III) were classified according to the Global Initiative for Chronic Obstructive Lung Disease guidelines (GOLD, 2011).
Period: Overall Study
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I - III)
Started | 20 | 23 | 29 | 20 | 34
Completed | 5 | 13 | 6 | 3 | 21
Not Completed | 15 | 10 | 23 | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Healthy Smokers: The healthy smoking group consisted of 20 current smokers with no history of respiratory disease
- Total: Total of all reporting groups
Arm/Group | Normal Subjects | Healthy Smokers | Mild-moderate Asthma | Severe Asthma | COPD (Gold Stage I - III) | Total
Number analyzed (Participants) | 29 | 20 | 20 | 23 | 34 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15) | 55 (10) | 41 (15) | 50 (14) | 66 (7) | 54 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 13 | 6 | 16 | 58
  Male | 15 | 11 | 7 | 17 | 18 | 68
Height [Mean (Standard Deviation); unit: centimeters] | 168.2 (10.7) | 167.2 (11.3) | 174.3 (10.1) | 168.7 (8.5) | 164.4 (8.5) | 168.1 (10.1)
Weight [Mean (Standard Deviation); unit: kilogram] | 73.05 (17.99) | 66.95 (15.55) | 76.30 (17.19) | 76.00 (13.18) | 69.75 (14.04) | 72.2 (15.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.63 (4.80) | 23.90 (4.82) | 24.90 (4.04) | 26.89 (5.64) | 25.76 (4.57) | 25.5 (4.8)
Smoking status [Number; unit: participants]
  Current smokers | 0 | 20 | 0 | 0 | 10 | 30
  Ex-smokers | 0 | 0 | 3 | 1 | 22 | 26

OUTCOME MEASURES:

1. Primary Outcome: FEV1
Description: Forced expiratory volume in one second
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: L
Groups:
- COPD (Gold Stage I-III): COPD patients (stages I - III) were classified according to the Global Initiative for Chronic Obstructive Lung Disease guidelines (GOLD, 2011).
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I-III)
Number analyzed (Participants) | 20 | 23 | 29 | 20 | 34
L | 3.03 (0.80) | 2.32 (0.88) | 3.18 (0.79) | 2.76 (0.73) | 1.67 (0.44)

2. Secondary Outcome: Calv
Description: Nitric oxide arising from the alveolar compartment.
Time Frame: 120 minutes
Measure: Mean (Standard Error); unit: ppb
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I - III)
Number analyzed (Participants) | 20 | 23 | 29 | 20 | 34
ppb | 4.3 (3.6) | 3.8 (3.2) | 2.9 (1.7) | 4.6 (2.9) | 3.7 (2.6)

3. Secondary Outcome: AX
Description: Reactance area for whole-breath
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I - III)
Number analyzed (Participants) | 20 | 23 | 29 | 20 | 34
kPa/L | 1.03 (1.05) | 1.88 (2.20) | 0.55 (0.57) | 0.82 (0.93) | 2.48 (2.12)

4. Secondary Outcome: R5 EX
Description: Resistance measured at 5 hertz during expiration
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: kPa/L/s
Groups:
- COPD (Gold Stage I - III): 1357
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I - III)
Number analyzed (Participants) | 20 | 23 | 29 | 20 | 34
kPa/L/s | 0.50 (0.17) | 0.60 (0.21) | 0.45 (0.16) | 0.50 (0.25) | 0.66 (0.24)

5. Secondary Outcome: J'aw
Description: Bronchial nitric oxide flux
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: nl/s
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I - III)
Number analyzed (Participants) | 20 | 23 | 29 | 20 | 34
nl/s | 138.5 (85) | 77.2 (62.4) | 76.2 (46.1) | 35.4 (21.2) | 60.7 (47.6)

6. Secondary Outcome: Sacin
Description: Ventilation heterogeneity within the acinar airways
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: /L
Arm/Group | Mild-moderate Asthma | Severe Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I-III)
Number analyzed (Participants) | 20 | 23 | 29 | 20 | 34
/L | 0.122 (0.094) | 0.214 (0.194) | 0.089 (0.051) | 0.150 (0.084) | 0.346 (0.139)

7. Secondary Outcome: Scond
Description: Ventilation heterogeneity within the conducting airways
Time Frame: 120 minutes
Population: Not all subjects have results for this parameter which is why the total number of results will not equal the number of participants recruited.
Measure: Mean (Standard Deviation); unit: /L
Arm/Group | Normal Subjects | Healthy Smokers | Mild-moderate Asthma | Severe Asthma | COPD (Gold Stage I - III)
Number analyzed (Participants) | 27 | 20 | 16 | 22 | 32
/L | 0.041 (0.016) | 0.068 (0.027) | 0.045 (0.015) | 0.057 (0.026) | 0.057 (0.020)

ADVERSE EVENTS:
Groups:
- Mild-moderate Asthma: Mild-moderate asthma recruited at baseline
- Sever Asthma: Sever Asthma recruited at baseline
- Normal Subjects: Normal subjects at baseline
- Healthy Smokers: Healthy smokers at baseline
- COPD (Gold Stage I - III): COPD (Gold stage I - III) baseline
Arm/Group | Mild-moderate Asthma | Sever Asthma | Normal Subjects | Healthy Smokers | COPD (Gold Stage I - III)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23 | 0/29 | 0/20 | 0/34
Other Adverse Events (participants affected / at risk) | 0/20 | 0/23 | 0/29 | 0/20 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes